CLINICAL TRIAL: NCT03559790
Title: Treatment Efficacy and Safety of Tenofovir Alafenamide (TAF) Switch Therapy in Patients Who Have Been Treated With Tenofovir Disoproxil Fumarate (TDF) in naïve Chronic Hepatitis B: a Real Life Multicenter Cohort Study in Korea
Brief Title: Treatment Efficacy and Safety of TDF-TAF Switch Study in South Korea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Myeong Jun Song, Associate Professor, The Catholic University of Korea
Other Study IDs: Gilead IN-US-320-4407
Record Dates: First submitted 2018-05-14; First posted 2018-06-18 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis b
Keywords: chronic hepatitis B; tenofovir alafenamide; tenofovir disoproxil fumarate; Safety; Efficacy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: tenofovir alafenamide — To evaluate of efficacy and safety in patients with TDF-TAF switch therapy

SUMMARY:
Recent TAF has introduced to have more safe profiles than TDF in clinical trials. Especially, TDF has the renal safety issue in high risk group including HIV, decompensated cirrhosis (ascites), uncontrolled DM etc.

However, there is no available cohort data for treatment efficacy and safety in TDF-TAF switch therapy in treatment-naïve chronic hepatitis B.

The aim of this study is to evaluate safety and efficacy of TAF switch therapy in patients with chronic hepatitis B who have been treated with TDF.

ELIGIBILITY:
Inclusion Criteria:

1. Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
2. Adult male and non-pregnant, non-lactating female subjects, 18 years of age and older, based on the date of the screening visit. A negative serum pregnancy test at Screening is required for female subjects of childbearing potential (unless surgically sterile or greater than 2 years post-menopausal).
3. Documented evidence of chronic HBV infection (e.g. HBsAg positive for more than 6 months)
4. Previous TDF naïve treatment (more than 96 weeks) baseline status including chronic hepatitis B with the following:

   * HBeAg-positive and HBeAb negative at Screening
   * Screening HBV DNA ≥ 1x 105 copies/mL
   * Screening serum ALT level ≥2×ULN(80 IU/L) and ≤ 10 ×ULN (by center laboratory range) OR
   * HBeAg-negative and HBeAb positive at Screening
   * Screening HBV DNA ≥ 1x 104 copies/mL
   * Screening serum ALT level ≥2×ULN(80 IU/L) and ≤ 10 ×ULN (by center laboratory range) OR
   * Cirrhosis at Screening
   * Screening HBV DNA ≥ 1x 104 copies/mL regardless of HBeAg status

     * Treatment naïve subjects defined as no history of antiviral therapy or < 12 weeks of oral antiviral treatment with any nucleoside or nucleotide analogue, including lamivudine or adefovir, clevudine, telbivudine, entecavir
5. The decision is made by the provider and patient to switch from TDF to TAF prior to discussion of the study of enrollment
6. Following the decision to switch therapy, signed written informed consent after being instructed about the objective and procedure of the clinical study
7. Must be willing and able to comply with all study requirements

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in the study.

1. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study.
2. Co-infection with HCV, HIV
3. Evidence of hepatocellular carcinoma (e.g. α-fetoprotein> 50 ng/mL or as evidenced by recent ultrasound or other standard of care measure)
4. Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible
5. Current alcohol or substance abuse judged by the investigator to potentially interfere with subject compliance
6. Currently receiving therapy with cytotoxic agent, nephrotoxic agents, or agents capable of modifying renal excretion
7. Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population that receive TDF-TAF switch therapy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Complete Virological response | at Week 96.
  Portion of subjects with plasma HBV DNA levels below 116 copies/mL
Incidence of of elevation of serum creatinine as a measure of renal safety | at Week 96
  Incidence of elevation of serum creatinine (>0.5mg/dL) from baseline creatinine
Incidence of osteopenia and osteoporosis as a measure of bone safety | at Week 96
  Incidence of osteopenia and osteoporosis according to Bone Mineral Density

SECONDARY OUTCOMES:
Biochemical response | at Week 48 and 96
  ALT normalization (Male <30 IU/L, Female <19 IU/L)
Serologic response | at Week 48 and 96
  loss rate of HBeAg in HBeAg positive patients
Serologic response | at Week 48 and 96
  seroconversion rate in HBeAg positive patients
Incidence of treatment-emergent adverse events | at Week 48 and 96
  all adverse events during tenofovir treatment

CONTACTS AND LOCATIONS:
Overall Officials: Myeong Jun Song, Principal Investigator — Daejeon St. Mary's hospital
Locations (1):
- The Catholic University of Korea, Daejeon St.Mary's Hosptial, Junggu, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No